CLINICAL TRIAL: NCT01172535
Title: A Phase II/III Trial of Lopinavir/Ritonavir Dosed According to the WHO Pediatric Weight Band Dosing Guidelines
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P1083; 10787 (Registry Identifier: DAIDS ES); IMPAACT P1083; NCT01338038 (obsolete NCT alias)
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2015-11

CONDITIONS: HIV
Keywords: Lopinavir/ritonavir; Pediatric dosing; World Health Organization
MeSH Terms: interventions — Lopinavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lopinavir/ritonavir (Experimental): Participants will receive lopinavir/ritonavir in addition to two nucleoside reverse transcriptase inhibitors (NRTIs) chosen by their doctors.
  Interventions: Drug: Lopinavir/ritonavir

INTERVENTIONS:
Drug: Lopinavir/ritonavir — Heat-stable tablets of 100 mg lopinavir, 25 mg ritonavir, or liquid formulation of 80 mg lopinavir, 20 mg ritonavir, dosed according to World Health Organization (WHO) pediatric weight band dosing guidelines
  Other Names: Kaletra; LPV/r

SUMMARY:
Treatment of children and infants with HIV requires modification of medication dosing according to a child's specific weight. For lopinavir/ritonavir (LPV/r), a second line treatment option that is increasingly necessary due to infant drug resistance, this dosing is often complicated and impractical in busy clinical settings. To address this, the World Health Organization (WHO) has released a simplified dosing table based on infant weight bands. This study will evaluate the absorption, safety, and tolerance of LPV/r in infants when dosed according to the new WHO guidelines.

DETAILED DESCRIPTION:
Because of previous exposure to nevirapine or other non-nucleoside reverse transcriptase inhibitors (NNRTIs), either by direct treatment or through their mothers in pregnancy, infants must often receive an alternate antiretroviral regimen that includes LPV/r. Dosing of LPV/r is currently based on a child's specific weight, and calculations of proper dosages are often too complicated to be practical in busy clinics, particularly those in limited resource settings. In order to simplify medication delivery and reduce prescribing errors, the WHO has released a dosing schedule for LPV/r based on groupings of infants and children by weight. This study will evaluate the pharmacokinetics, safety, and tolerance of LPV/r dosed according to these guidelines. The following strata were used to guide accrual:

Number of Participants to be Enrolled by Weight Band:

3-4.9 kg: 11 liquid

5-6.9 kg: 11 liquid

7-9.9 kg: 17 liquid

10-16.9 kg: 11 liquid, 22 tablet

17-19.9 kg: 11 tablet

20-24.9 kg: 11 tablet

Participation in this study will last 6 months. Infant participants and their caretakers will need to attend study visits at entry and Weeks 2, 4, 12, and 24. At entry, participants will be given LPV/r either in liquid or tablet form, depending on whether they can swallow pills. Dosing will be calculated using the WHO schedule. At all study visits, participants will undergo a physical exam and caretakers will be asked about how well the child is taking the study medications. In addition, at Weeks 4, 12, and 24, blood samples will be taken from the participant to determine health and levels of the medication in the body. The visit on Week 4 will also require pharmacokinetic testing, which means the child will need to be monitored at the hospital for 12 hours and complete six additional blood drawls. All other study visits will last 1 to 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Weight equal to or greater than 3 kg, but less than 25 kg, at the time of enrollment
* Confirmed diagnosis of HIV-1 infection
* Lopinavir/ritonavir (LPV/r)-treatment naïve and LPV/r-treatment eligible as defined by country-specific guidelines or the WHO pediatric treatment guidelines and confirmed by investigator
* Willingness to take two nucleoside reverse transcriptase inhibitos (NRTIs), in accordance with appropriate national or international treatment guidelines
* Demonstrated ability and willingness to swallow tablets for children larger than 10 kg. This can be assessed before inclusion (for example, a test trial with similar size solid tablet such as tic-tac).
* Participants in the weight band between 10 and 16.9 kg that are unable to swallow tablets will receive liquid formulation
* Parent or legal guardian able and willing to provide written informed consent

Exclusion Criteria:

* Planned concurrent use of non-nucleoside reverse transcriptase inhibitors (NNRTIs), integrase inhibitors, or an entry inhibitor
* Planned concurrent protease inhibitor (PI) use, other than LPV/r
* Prior treatment with LPV/r. Prior treatment with other PIs is allowed.
* Results of certain laboratory tests indicating adverse events of Grade 3 or greater
* Results of a lipase test indicating adverse event of Grade 2 or greater or clinical evidence of pancreatitis within 30 days prior to study entry
* Tuberculosis co-treatment with rifampicin-containing regimen
* Treatment with any enzyme-inducing antiepileptic drugs, such as henobarbital, phenytoin or carbamazepine
* Clinical condition requiring the use of a prohibited medication (see protocol for more details)
* Clinically unstable child requiring acute treatment for a serious opportunistic infection
* Chemotherapy for active malignancy
* Any clinically significant diseases (other than HIV-1 infection) or clinically significant findings during the screening medical history or physical examination that, in the investigator's opinion, would compromise participation in this study
* Treatment with experimental drugs for any indication within 30 days prior to study entry
* Known history of cardiac conduction abnormality and/or underlying structural heart disease, including congenital long QT

Min Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2010-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A. Pinto, MD, Study Chair — Federal University of Minas Gerais
Locations (19):
- United States (3):
  - University of California, UC San Diego CRS, La Jolla, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Boston Medical Center Ped. HIV Program NICHD CRS, Boston, Massachusetts
- Brazil (7):
  - SOM Federal University Minas Gerais Brazil NICHD CRS, Belo Horizonte, Minas Gerais
  - Hosp. Santa Casa Porto Alegre Brazil NICHD CRS, Porto Alegre, Rio Grande do Sul
  - Hospital Federal dos Servidores do Estado NICHD CRS, Rio de Janeiro
  - Instituto de Puericultura e Pediatria Martagao Gesteira - UFRJ NICHD CRS, Rio de Janeiro
  - Hosp. Geral De Nova Igaucu Brazil NICHD CRS, Rio de Janeiro
  - Inst de Infectologia Emilio Ribas Sao Paulo Brazil NICHD CRS, São Paulo
  - Univ. of Sao Paulo Brazil NICHD CRS, São Paulo
- South Africa (2):
  - Shandukani CRS, Johannesburg, Gauteng
  - Family Clinical Research Unit (FAM-CRU) CRS, Tygerberg, Western Cape
- Thailand (7):
  - Bhumibol Adulyadej Hosp. CRS, Saimai, Bangkok
  - Siriraj Hospital Mahidol University CRS, Bangkok, Bangkoknoi
  - Prapokklao Hosp. CRS, Chanthaburi
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai
  - Chiangrai Prachanukroh Hospital CRS, Chiangrai
  - Chonburi Hosp. CRS, Chon Buri
  - Phayao Provincial Hosp. CRS, Phayao

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 97 participants enrolled from 19 clinical sites in four countries. There were 57 participants on the liquid formulation and 40 on tablet. Accrual took place from May 20, 2011 through June 19, 2013.
Pre-assignment Details: HIV-infected infants and children ≥3 to <25 kg had to be LPV/r-treatment naïve. Children ≥10 kg had to demonstrate ability and willingness to swallow tablets. Participants were stratified by weight and drug formulation (liquid vs. tablet).
Groups:
- Lopinavir/Ritonavir: Participants receiving lopinavir/ritonavir, dosed according to World Health Organization (WHO) pediatric weight band dosing guidelines, in addition to two nucleoside reverse transcriptase inhibitors (NRTIs) chosen by their doctors.
Period: Overall Study
Arm/Group | Lopinavir/Ritonavir
Started | 97
Completed | 89
Not Completed | 8
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Ineligible at study entry | 1
Not completed — Unwilling to adhere to study requirement | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled in the study
Groups:
- Lopinavir/Ritonavir: Participants receiving lopinavir/ritonavirr, dosed according to World Health Organization (WHO) pediatric weight band dosing guidelines, in addition to two nucleoside reverse transcriptase inhibitors (NRTIs) chosen by their doctors.
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 97
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 2.5 [0.5 to 6.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 37
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 39
  White | 7
  More than one race | 0
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  United States | 5
  Brazil | 32
  South Africa | 23
  Thailand | 37
HIV RNA (copies/mL) at study entry [Median (Inter-Quartile Range); unit: log copies/mL] | 5.2 [4.6 to 5.7]
CD4% at study entry [Median (Inter-Quartile Range); unit: percentage of total lymphocytes] | 24.2 [15.8 to 29.0]

OUTCOME MEASURES:

1. Primary Outcome: Lopinovir/Ritonavir Area Under the Concentration-time Curve (AUC0-24)
Description: Area under the curve over 24 hours (AUC0-24), as determined by a non-compartmental analysis of 12-hour pharmacokinetic sampling for lopinavir/ritonavir
Time Frame: Measured at 4 weeks of treatment prior to the observed dose and at 2, 4, 6, 8, and 12 hours post-dose
Population: Participants having complete pharmacokinetics data at week 4
Measure: Geometric Mean (90% Confidence Interval); unit: mcg*hr/mL
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 81
mcg*hr/mL | 196 [177 to 217]

2. Primary Outcome: Maximum Concentration of Lopinavir/Ritonavir (Cmax)
Description: Maximum concentration of lopinavir/ritonavir, as determined by analysis of 12-hour pharmacokinetic sampling
Time Frame: Measured at 4 weeks of treatment prior to the observed dose and at 2, 4, 6, 8, and 12 hours post-dose
Population: Participants having complete pharmacokinetics data at week 4
Measure: Geometric Mean (90% Confidence Interval); unit: mcg/mL
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 81
mcg/mL | 11.25 [10.24 to 12.35]

3. Primary Outcome: Minimum Concentration of Lopinavir/Ritonavir (Cmin)
Description: Minimum concentration of lopinavir/ritonavir, as determined by analysis of 12-hour pharmacokinetic sampling
Time Frame: Measured at 4 weeks of treatment prior to the observed dose and at 2, 4, 6, 8, and 12 hours post-dose
Population: Participants having complete pharmacokinetics data at week 4
Measure: Geometric Mean (90% Confidence Interval); unit: mcg/mL
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 81
mcg/mL | 2.47 [1.52 to 4.02]

4. Primary Outcome: Clearance of Lopinavir/Ritonavir (CL/F)
Description: Clearance of lopinavir/ritonavir, as determined by analysis of 12-hour pharmacokinetic sampling
Time Frame: Measured at 4 weeks of treatment prior to the observed dose and at 2, 4, 6, 8, and 12 hours post-dose
Population: Participants having complete pharmacokinetics data at week 4
Measure: Geometric Mean (90% Confidence Interval); unit: L/h/kg
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 81
L/h/kg | 0.15 [0.13 to 0.17]

5. Primary Outcome: Proportion of Participants With an AUC of Less Than 10% of Adults
Description: Proportion of participants with an AUC less that 10% of adults (AUC0-24 <104 mcg*hr/mL)
Time Frame: Measured at 4 weeks of treatment prior to the observed dose and at 2, 4, 6, 8, and 12 hours post-dose
Population: Participants with complete pharmacokinetics data at week 4
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 81
proportion of participants | 0.15 [0.09 to 0.23]

6. Secondary Outcome: Adherence
Description: Adherence, defined as proportion of doses taken (note: proportion could be greater than 1.0 for reasons such as tablets having to be taken twice due to first one being spit out or imprecise measurement of liquid doses)
Time Frame: Measured at week 4, week 12, and study completion (week 24)
Population: Participants bringing medication to be measured at the study visit
Measure: Median (Inter-Quartile Range); unit: Proportion of expected doses taken
Groups:
- Week 4: Participants bringing medication to be measured at study week 4
- Week 12: Participants bringing medication to be measured at study week 12
- Week 24: Participants bringing medication to be measured at study week 24
Arm/Group | Week 4 | Week 12 | Week 24
Number analyzed (Participants) | 62 | 59 | 59
Proportion of expected doses taken | 1.00 [0.97 to 1.10] | 0.99 [0.88 to 1.01] | 1.00 [0.91 to 1.01]

7. Secondary Outcome: Treatment Efficacy (HIV Viral Load)
Description: Having HIV viral load <400 copies/mL at the week 24 visit
Time Frame: Measured at entry and study completion (week 24)
Population: Participants with data from both study entry and the week 24 study visit
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 79
proportion of participants | 0.72 [0.61 to 0.82]

8. Secondary Outcome: Treatment Efficacy (CD4%)
Description: Having CD4%≥25 at the week 24 visit.
Time Frame: Measured at entry and study completion (week 24)
Population: Participants with data from both study entry and the week 24 study visit
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 83
proportion of participants | 0.71 [0.60 to 0.81]

9. Primary Outcome: Number of Participants Experiencing Adverse Events of Grade 3 or 4
Description: Adverse events were graded by the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, dated December, 2004, Clarification August 2009, which is available on the RSC web site (http://rsc.tech-res.com/safetyandpharmacovigilance/). Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = potentially life-threatening, Grade 5 = death
Time Frame: Measured at study visits through end of study (weeks 2, 4, 12, 24)
Population: All participants
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 97
participants | 32

10. Primary Outcome: Proportion of Participants Tolerating LPV/r
Description: Participants were considered to have tolerated medication if they did not stop treatment before the 24 week PK visit for any reason other than completing treatment or death not related to treatment.
Time Frame: Measured at study completion (week 24)
Population: All participants
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Lopinavir/Ritonavir
Number analyzed (Participants) | 97
proportion of participants | 0.93 [0.86 to 0.97]

ADVERSE EVENTS:
Time Frame: From entry until off-study (week 24)
Description: Expedited adverse event (AE) reporting followed Intensive Division of AIDS (DAIDS) Reporting Level, which included Aes resulting in death, significant disabilities, requiring hospitalization, and ≥grade 3 Aes defined by the "DAIDS Table for Grading the Severity of Adult and Pediatric Aes", V1.0, 12/2004.
Groups:
- LPV/r: Participants receiving lopinavir/ritonavir, dosed according to World Health Organization (WHO) pediatric weight band dosing guidelines, in addition to two nucleoside reverse transcriptase inhibitors (NRTIs) chosen by their doctors.
Arm/Group | LPV/r
Serious Adverse Events (participants affected / at risk) | 20/97
Other Adverse Events (participants affected / at risk) | 96/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LPV/r (N=97)
Neutropenia (Blood and lymphatic system disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Drowning (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 1
Immune reconstitution inflammatory syndrome associated tuberculosis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Measles (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 6
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1
Amylase increased (Investigations) | 3
Hyperamylasaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LPV/r (N=97)
Lymphadenopathy (Blood and lymphatic system disorders) | 8
Conjunctival pallor (Eye disorders) | 5
Eye discharge (Eye disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 33
Vomiting (Gastrointestinal disorders) | 30
Pyrexia (General disorders) | 42
Hepatomegaly (Hepatobiliary disorders) | 9
Immune reconstitution inflammatory syndrome (Immune system disorders) | 5
Bronchitis (Infections and infestations) | 6
Gastroenteritis (Infections and infestations) | 13
Impetigo (Infections and infestations) | 7
Oral candidiasis (Infections and infestations) | 6
Pharyngitis (Infections and infestations) | 6
Pneumonia bacterial (Infections and infestations) | 7
Alanine aminotransferase abnormal (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 18
Amylase abnormal (Investigations) | 39
Aspartate aminotransferase increased (Investigations) | 18
Blood bicarbonate decreased (Investigations) | 54
Blood calcium decreased (Investigations) | 11
Blood calcium increased (Investigations) | 25
Blood cholesterol increased (Investigations) | 19
Blood glucose decreased (Investigations) | 19
Blood glucose increased (Investigations) | 9
Blood magnesium decreased (Investigations) | 10
Blood phosphorus decreased (Investigations) | 8
Blood potassium decreased (Investigations) | 7
Blood potassium increased (Investigations) | 14
Blood sodium decreased (Investigations) | 58
Breath sounds abnormal (Investigations) | 7
Haemoglobin decreased (Investigations) | 40
Neutrophil count decreased (Investigations) | 25
Platelet count decreased (Investigations) | 7
Decreased appetite (Metabolism and nutrition disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 48
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12
Rales (Respiratory, thoracic and mediastinal disorders) | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 43
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 11
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 6
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 6
Papule (Skin and subcutaneous tissue disorders) | 13
Rash (Skin and subcutaneous tissue disorders) | 18
Skin exfoliation (Skin and subcutaneous tissue disorders) | 6
Skin lesion (Skin and subcutaneous tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and seven (7) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights